CLINICAL TRIAL: NCT04490525
Title: Future Patient - Telerehabilitering af Patienter Med Hjertesvigt II
Brief Title: Future Patient - Telerehabilitation of Patients With Heart Failure II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Aage and Johanne Louis-Hansens Foundation (Unknown); Laboratory of Welfare Technology, Department of Health Science and Technology, AAU (Unknown); Viborg Regional Hospital (Other); Skive Healthcare Center (Unknown); Viborg Healthcare Center (Unknown); University of Aarhus (Other); Department of Photonics Engineering, Technical University of Denmark (Unknown)
Responsible Party: Principal Investigator, Birthe Dinesen, Professor, PhD, Master in Political Science, RN, Head of Laboratory of Welfare Technology - Telehealth & Telerehabilitation, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20200037
Record Dates: First submitted 2020-07-19; First posted 2020-07-29 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will participate in the telerehabilitation program (please see detailed description of telerehabilitation program and technologies). The two steps in the telerehabilitation program last up to six months depending on how fast the titration of medicine in step one will be conducted. The intervention group will spend 5-10 minutes every day on monitoring themselves. Every month, an online questionnaire has to be filled in which will take up to 5 minutes. At enrolment, after titration of medicine, and the end of rehabilitation, the patient will fill in an online questionnaire. This will take 5 minutes each time. Selected patients and relatives will be asked if they wish to participate in interviews after participation in the trial. Each interview will last less than one hour. Number of interviews will be decided when data saturation has been achieved.
  Interventions: Device: Telerehabilitation
- Control (No Intervention): The control group will follow a conventional rehabilitation program (Egstrup et al 2015). The control subjects will participate in medicine titration for 1- 3 months and conventional rehabilitation for 3 months. The participation in the control group will last up to six months. The exact period depends on how fast the titration of medicine is conducted. At enrolment, after titration of medicine, and end of rehabilitation, the patient will fill in a questionnaire. This will take 5 minutes each time.

INTERVENTIONS:
Device: Telerehabilitation — Blood pressure (iHealth Neo/BP5s), weight (iHealth Lina), step counters(Fitbit Inspire & Charge 3), sleep sensor (Emfit QS), and tablet (iPad Air 2).
  Arms: Intervention

SUMMARY:
The aim of the study is to test and evaluate the use of video consultations and an algorithm for weight gain and loss in the Future Patient Telerehabilitation program for HF patients in an RCT.

DETAILED DESCRIPTION:
Next steps The Future Patient study - telerehabilitation of HF patients II

Based on the preliminary results from FP I (being published fall 2020) and a review of literature, the investigators would like to improve our telerehabilitation program and technologies in order to prepare for implementation of the FTP and technologies.

* The HF patients in FP I expressed that the KCCQ was too long when having to complete the questionnaire every other week. Therefore, the investigators would like to test a shorter questionnaire HeartQoL (ESC) as a patient-reported outcome tool every month.
* Video consultations instead of physical meetings with doctors and nurses at the hospital. Currently, there is a lack of evidence regarding the use of video to decrease physical visits at the hospitals instead of video consultations.
* Test of algorithms for detecting an increase in weight on two days following clinical cardiac guidelines (Ponikowski et al 2016).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HF NYHA Class II-IV, who have a current hospitalization for acute decompensated HF or a visit to the HF outpatient clinic within the past two weeks
* Patients with an EF of 40% or less
* Adults (18 years or older); no upper age limit
* Patients living in Viborg and Skive Municipality
* Patients living at home and capable of caring for themselves
* Have basic computer skills or a relative who have basic computer skills

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present and previous neurologic, musculoskeletal or cognitive disability or active psychiatric history (as noted in the medical record) other than depression or anxiety related to cardiac or other chronic illness
* Lack of ability to cooperate
* Does not speak/read/understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Intervention: at baseline, after 1 month, after 2 months, after 3 months, after 4 months, after 5 months, after 6 months. Control: baseline, after 3 months, after 6 months
  15 % increase in health-related quality of life measured by HeartQoL

SECONDARY OUTCOMES:
Reduction of the number of visits to the outpatient clinic | For both intervention and control group: 6 months
  Number of visits to the outpatient clinic between intervention and control group
Number of readmissions | For both intervention and control group: 6 months
  Number of readmissions between intervention and control group
Number of tele-communicational (phone and video) contacts | For both intervention and control group: 6 months
  Number of phone and video contacts to the healthcare professionals between intervention and control group
Experiences of HF patients and healthcare professionals with the use of video consultations | Intervention group: at month 6
  Interviews with HF patients and healthcare professionals regrind their experiences with the use of video consultations
Testing an algorithm on weight based on adherence | Intervention group: at baseline, week: 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
  Questionnaires about feedback from an algorithm on weight
Degree of depression | For both intervention and control group: at baseline, 3 months, and 6 months
  Degree of depression measured through HADS questionnaire
Use of the website "Hjerteportalen.dk" | Intervention group: 6 months
  Use of the website "Hjerteportalen.dk" based on log files

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Viborg Regional Hospital, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Read about project — https://www.labwelfaretech.com/en/